CLINICAL TRIAL: NCT04225533
Title: SP16 Inflammatory Response Inhibition Trial
Acronym: SPIRIT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Serpin Pharma, LLC (Other)
Collaborators: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HM20018201
Record Dates: First submitted 2020-01-08; First posted 2020-01-13 (Actual); Results first posted 2023-01-30 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Myocardial Infarction; Inflammation
MeSH Terms: conditions — Myocardial Infarction; Inflammation

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SP16 (Experimental): Patients will receive a single dose of SP16 0.2 mg/kg by subcutaneous injection
  Interventions: Drug: SP16

INTERVENTIONS:
Drug: SP16 — All patients will receive a single dose of SP16

SUMMARY:
This study will evaluate the potential benefit of blocking inflammation during a heart attack using an investigational anti-inflammatory medicine called SP16. The study will enroll 10 patients and all 10 patients will receive a standard dose of SP16.

DETAILED DESCRIPTION:
The main hypothesis of this study is that a single subcutaneous administration of SP16 0.2 mg/kg is safe and well tolerated in patients with ST segment elevation myocardial infarction (STEMI) and associated with a reduction in the acute inflammatory response to STEMI, as measured as area-under-the-curve (AUC) for C reactive protein (CRP), the preferred inflammatory marker for cardiovascular risk prognostication.

SP16 will be administered subcutaneously as this route has greater ease of administration than intravenous injection. A single dose administration has been selected based upon pre-clinical data and expected clinical use of SP16.

ELIGIBILITY:
In order to be eligible for this study, patients must meet all the 3 criteria:

1. Presentation to the hospital with acute STEMI defined as chest pain (or equivalent) with an onset within 12 hours and electrocardiogram (ECG) evidence of ST segment elevation (>1 mm) in 2 or more anatomically contiguous leads that is new or presumably new (for intermittent pain lasting more than 12 hours, the time from the when the pain became severe and constant);
2. Coronary intervention planned and/or completed within 12 hours of symptom onset, and enrollment in the study within 6 hours of angiogram (max 18 hours from symptom onset)
3. Age>21 years

In order to be eligible for this study, patients must meet none of the Exclusion criteria.

* Inability to give informed consent
* Hemodynamic instability as defined as need for inotropic or vasoactive agents, or need for mechanical support devices (including intra-aortic balloon pump)
* Pregnancy or breastfeeding
* Preexisting congestive heart failure (American Heart Association/American College of Cardiology class C-D, New York Heart Association III-IV)
* Preexisting severe left ventricular dysfunction (LVEF<20%)
* Preexisting severe valvular heart disease
* Known active infections (acute or chronic)
* Recent (<14 days) or active use of immunosuppressive drugs (including but not limited to high-dose corticosteroids [>1 mg/kg of prednisone equivalent], tumor necrosis factor-alpha blockers, cyclosporine) not including non-steroidal anti-inflammatory drugs (NSAIDs) or corticosteroids used for intravenous (IV) dye allergy only)
* Recent (<14 days) or active use of anti-inflammatory drugs (not including NSAIDs or corticosteroids used for IV dye allergy only)
* Known chronic inflammatory disease (including but not limited to rheumatoid arthritis, systemic lupus erythematosus)
* Known active malignancy of any type, or prior diagnosis in the past 10 years
* Neutropenia (absolute neutrophil count<1,800/mm3 [or <1,000/mm3 in African American patients])
* Severe impairment in renal function (estimated glomerular filtration rate <30 ml/kg*min)
* Anticipated need for cardiac or major surgery
* Known Allergy to SP16

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-02-24 (Actual); Primary Completion 2021-01-04 (Actual); Study Completion 2021-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Abbate, MD, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Van Tassell BW, Wohlford GF, Del Buono MG, Damonte JI, Markley R, Turlington J, Kadariya D, Talasaz A, Ho J, Marawan A, Thomas GK, Austin D, Gineste C, Gelber C, Abbate A. Safety, Tolerability, and Effects of a Single Subcutaneous Administration of SP16 - a SERPIN-like, Small Peptide Agonist of the Low-Density Lipoprotein-like Receptor 1- on the Acute Inflammatory Response in Patients With ST-Segment Elevation Myocardial Infarction. J Cardiovasc Pharmacol. 2022 Nov 1;80(5):672-678. doi: 10.1097/FJC.0000000000001331. PMID 35881895

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SP16
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | SP16
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 55 [51 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve (AUC) for C-reactive Protein (CRP)
Description: This study will evaluate the anti-inflammatory effect of SP16 by calculating the AUC for CRP. This is done by measuring CRP at baseline, 72 hours, and 14 days. The AUC will then be compared to historical controls to evaluate whether or not SP16 reduces the AUC for CRP.
Time Frame: Baseline, 72 hours, 14 days
Measure: Median (Inter-Quartile Range); unit: mg*day/L
Arm/Group | SP16
Number analyzed (Participants) | 10
mg*day/L | 133 [46 to 528]

2. Secondary Outcome: Area Under Curve (AUC) for Creatine-Kinase Myocardial Band (CK-MB)
Description: This study will estimate the infarct size based upon area under the curve (AUC) for creatine-kinase myocardial band (CK-MB). The AUC calculation will come from CK-MB levels drawn during usual care. The infarct size will then be compared to historical controls to evaluate whether or not SP16 reduces the infarct size.
Time Frame: 72 hours
Measure: Median (Inter-Quartile Range); unit: ng/mL*day
Arm/Group | SP16
Number analyzed (Participants) | 10
ng/mL*day | 1432 [675 to 3089]

3. Secondary Outcome: Change in Left Ventricular Ejection Fraction (LVEF) at Baseline and 365 Days
Description: Patients will undergo transthoracic echocardiography at baseline and 365 days to evaluate the change in LVEF.
Time Frame: 365 days
Measure: Median (Inter-Quartile Range); unit: percentage of LVEF
Arm/Group | SP16
Number analyzed (Participants) | 8
percentage of LVEF | 5 [-0.6 to 9]

4. Secondary Outcome: Diagnosis of Heart Failure
Description: Number of participants diagnosed with heart failure at 1 year follow up
Time Frame: 365 days
Measure: Count of Participants; unit: Participants
Arm/Group | SP16
Number analyzed (Participants) | 10
Participants | 0

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | SP16
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 2/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SP16 (N=10)
Cardiac disorders (Cardiac disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI shall be free to publish and/or present about the Study. All publications must be submitted to the sponsor at least 30 days prior to submission for review/comment. PI will consider any such comments in good faith but is under no obligation to incorporate. If Sponsor notifies PI that it desires patent applications, PI will defer Publication for a period not to exceed 60 days; & if Publication contains Company's Confidential, the PI agrees to delete such Company's Confidential Information.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-21): https://cdn.clinicaltrials.gov/large-docs/33/NCT04225533/Prot_SAP_000.pdf